CLINICAL TRIAL: NCT01110005
Title: A Multi-Center, Two-Arm, Single-Blind Randomized Trial of IV Fluids During Labor
Brief Title: A Trial of Intravenous Fluids During Labor
Acronym: RARHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Lehigh Valley Hospital (Other); The Reading Hospital and Medical Center (Other); St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32118
Record Dates: First submitted 2010-04-09; First posted 2010-04-23 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2017-01

CONDITIONS: Ketosis
Keywords: D5LR; glucose containing IV solution; LR; non glucose IV solution
MeSH Terms: conditions — Ketosis | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D5 Lactated Ringer's solution (D5LR) (Active Comparator): IV fluid containing glucose administered throughout labor at an average infusion rate of 125 ml/hr.
  Interventions: Other: D5 Lactated Ringer's Solution (D5LR)
- Lactated Ringer's solution (LR) (Active Comparator): Non-glucose IV fluid administered throughout labor at an average infusion rate of 125 ml/hr.
  Interventions: Other: Lactated Ringer's Solution (LR)

INTERVENTIONS:
Other: D5 Lactated Ringer's Solution (D5LR) — D5LR IV fluid
  Arms: D5 Lactated Ringer's solution (D5LR)
Other: Lactated Ringer's Solution (LR) — LR IV fluid
  Arms: Lactated Ringer's solution (LR)

SUMMARY:
The purpose of this study is to determine if intrapartum use of a glucose-containing solution will improve the outcomes in pregnant women and their babies.

DETAILED DESCRIPTION:
This will be a multi-center, prospective, single-blind randomized trial of two types of IV fluids for maintenance hydration during labor. This study will be conducted at 4 sites: Reading (Reading Hospital), Allentown (Lehigh Valley), St. Luke Hospital and Hershey (Penn State College of Medicine). It will include 1524 pregnant women at ≥ 36 weeks presenting in spontaneous labor for anticipated delivery.

The primary research hypothesis is that intravenous hydration during labor with a glucose-containing fluid will lead to more efficient uterine contractility and will lead to a reduction of cesarean delivery. The primary outcome measure is the occurrence of a cesarean birth during the study period. The primary analysis will use an intent-to-treat approach to examine differences between the two IV fluid treatments in the proportion of deliveries requiring cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Women of any age with a singleton gestation in spontaneous labor at greater than or equal to 36 weeks without contraindication to participation.
2. These women will be in good health and candidates for vaginal delivery.

Exclusion Criteria:

1. Patients who are not candidates for vaginal delivery. This may be due to fetal malpresentation, prior cesarean section, multiple gestations, etc.
2. Patients presenting for induction of labor or requiring induction upon admission.
3. Patients presenting for scheduled cesarean section.
4. Patients with any form of diabetes or glucose dysregulation condition.
5. Concurrent use of steroids.
6. Patients presenting in active labor with advanced cervical dilation (≥ 6 cm).
7. Subjects participating in another labor and delivery related clinical trial that conflicts with this trial (as determined by the site PI).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Study Director — The Pennsylvania State University College of Medicine, Hershey, Pennsylvania, United States; John Smulian, M.D., Principal Investigator — Lehigh Valley Hospital, Allentown, Pennsylvania, United States
Locations (4):
- United States (4):
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke Hospital, Bethlehem, Pennsylvania
  - The Penn State University, Hershey, Pennsylvania
  - The Reading Hospital and Medical Center, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dapuzzo-Argiriou LM, Smulian JC, Rochon ML, Galdi L, Kissling JM, Schnatz PF, Gonzalez Rios A, Airoldi J, Carrillo MA, Maines J, Kunselman AR, Repke J, Legro RS. A multi-center randomized trial of two different intravenous fluids during labor. J Matern Fetal Neonatal Med. 2016;29(2):191-6. doi: 10.3109/14767058.2014.998190. Epub 2015 Sep 4. PMID 25758624

RESULTS

PARTICIPANT FLOW:
Groups:
- D5 Lactated Ringers Solution (D5LR): IV fluid containing glucose administered throughout labor at an average infusion rate of 125 ml/hr.
- Lactated Ringers Solution (LR): Non-glucose IV fluid administered throughout labor at an average infusion rate of 125 ml/hr.
Period: Overall Study
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR)
Started | 157 | 161
Completed | 153 | 156
Not Completed | 4 | 5
Not completed — ineligible | 1 | 2
Not completed — missing consent | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 318 subjects were randomized for the study but nine were excluded from analysis entirely: 3 were deemed ineligible, 5 did not have adequate documentation of informed consent, and 1 subject withdrew consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR) | Total
Number analyzed (Participants) | 153 | 156 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (4.9) | 26.8 (4.9) | 26.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 156 | 309
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 12 | 33
  Not Hispanic or Latino | 131 | 144 | 275
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 129 | 127 | 256
  African American | 4 | 11 | 15
  Other | 18 | 18 | 36
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: C-Section
Description: Compare c-section rates between the D5LR and LR treatment groups
Time Frame: From onset of labor to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR)
Number analyzed (Participants) | 153 | 156
Participants | 23 | 18
Statistical Analysis 1: Comparison: D5 Lactated Ringers Solution (D5LR) vs Lactated Ringers Solution (LR); Test type: Superiority; p = 0.34, Regression, log binomial; The regression model adjusted for site of recruitment as a covariate; Risk Ratio (RR) = 1.3, 95% CI 2-sided [0.7 to 2.3] — D5LR vs. LR

2. Secondary Outcome: Oxytocin Augmentation
Description: Compare augmentation rates between the D5LR and LR treatment groups
Time Frame: From onset of labor to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR)
Number analyzed (Participants) | 153 | 156
Participants | 92 | 88
Statistical Analysis 1: Comparison: D5 Lactated Ringers Solution (D5LR) vs Lactated Ringers Solution (LR); Test type: Superiority; p = 0.40, Regression, log binomial; The regression model adjusted for site of recruitment as a covariate; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.9 to 1.3] — D5LR vs. LR

3. Secondary Outcome: Time to Delivery
Description: Compare time to delivery between the D5LR and LR treatment groups
Time Frame: From onset of labor to delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR)
Number analyzed (Participants) | 150 | 150
hours | 12.8 [7.6 to 18.3] | 12.1 [8.4 to 18.0]
Statistical Analysis 1: Comparison: D5 Lactated Ringers Solution (D5LR) vs Lactated Ringers Solution (LR); Test type: Superiority; p = 0.69, Cochran-Mantel-Haenszel; This method was used to control for site of recruitment

ADVERSE EVENTS:
Time Frame: From onset of labor through the mother's hospital stay
Description: Adverse event information was collected via review of medical charts.
Arm/Group | D5 Lactated Ringers Solution (D5LR) | Lactated Ringers Solution (LR)
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/156
Serious Adverse Events (participants affected / at risk) | 1/153 | 5/156
Other Adverse Events (participants affected / at risk) | 2/153 | 9/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D5 Lactated Ringers Solution (D5LR) (N=153) | Lactated Ringers Solution (LR) (N=156)
Congenital anomalies (General disorders) | 1 (1) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | D5 Lactated Ringers Solution (D5LR) (N=153) | Lactated Ringers Solution (LR) (N=156)
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2/149 (2) | 9/151 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No